CLINICAL TRIAL: NCT04339283
Title: Standardized Hibiscus Sabdariffa Linn Tea, Potential Nutraceutical Candidate for the Prevention of Hypertension, Diabetes, and Hypercholesterolemia - a Pilot Study
Brief Title: Effect of Standardized Hibiscus Sabdariffa Tea in Seemingly Healthy Human Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ibadan (Other)
Responsible Party: Principal Investigator, SEGUN SHOWANDE, Dr., University of Ibadan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hibiscus-tea Study
Record Dates: First submitted 2020-03-31; First posted 2020-04-09 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Healthy Human Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standardized Hibiscus sabdariffa tea Arm (Experimental): 300 mL of freshly prepared standardized Hibiscus sabdariffa tea (containing 102.49 mg/L of total monomeric anthocyanin) is administered daily to the participants for 28 days
  Interventions: Dietary Supplement: Standardized Hibiscus sabdariffa tea
- Water Arm (No Intervention): 300 mL of distilled water is administered to the participants daily for 28 days.

INTERVENTIONS:
Dietary Supplement: Standardized Hibiscus sabdariffa tea — Daily consumption of Standardized Hibiscus sabdariffa tea
  Arms: Standardized Hibiscus sabdariffa tea Arm

SUMMARY:
Hibiscus sabdariffa tea is commonly used all over the world by healthy individual but the tea is also employed by patients in the management of chronic diseases such as hypertension diabetes, high cholesterol, liver disease etc. Several studies in humans and animal have proved the efficacy of Hibiscus sabdariffa tea in lowering blood pressure, blood glucose level and serum total cholesterol. But no study exists on the effect of daily consumption of this tea on blood pressure, blood glucose, total cholesterol and other biochemical and hematological parameters in healthy humans. Hence this study.

DETAILED DESCRIPTION:
Several studies have been carried out on the effect of the water beverage of Hibiscus sabdariffa, most focus on hypertensive patients, diabetic patients and obese patient and some studies investigated the hypolipidemic a effect of the water beverage of Hibiscus sabdariffa as well as its effect on haematological parameters but mice were used for these studies. Little or no investigation has been done to assess the safety of daily consumption of this water beverage of hibiscus sabdariffa on humans.

Hence, this study aims at investigating the safety in the daily consumption of Zobo in humans, monitoring lipid profile, blood pressure, blood glucose, body mass index and haematological parameters such as haematocrit, haemoglobin, total white blood cells and also hepatic indices.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers only
* Not on any medications or herbs
* No disease condition
* Females not pregnant
* Non-smokers

Exclusion Criteria:

* Below 18yrs or above 40 years
* presence of chronic disease
* on medications pregnant females

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Systolic Blood Pressure and Diastolic Blood Pressure on the 14th day | 14 days
  Blood pressure was measured in mmHg at baseline and on the 14th day of study with the aid of Omron Digital Blood pressure monitor
Change from Baseline Systolic Blood Pressure and Diastolic Blood Pressure on the 28th day | 28 days
  Systolic and Diastolic Blood pressures were measured in mmHg at baseline and on the 28th day of study with the aid of Omron Digital Blood pressure monitor
Change from Baseline Fasting Blood Glucose level on the 14th day | 14 days
  Fating blood glucose level was measured with AccuChek Active glucometer in mg/dL on the 14th day of study
Change from Baseline Fasting Blood Glucose level on the 28th day | 28 days
  Fating blood glucose level was measured with AccuChek Active glucometer in mg/dL on the 28th day of study
Change from Baseline Total Serum Cholesterol on the 14th day | 14 days
  Total Serum Cholesterol was analysed with Randox kit and measured in mg/dL on the 14th day
Change from Baseline Total Serum Cholesterol on the 28th day | 28 days
  Total Serum Cholesterol was analysed with Randox kit and measured in mg/dL on the 28th day
Change from Baseline Triglyceride on the 14th day | 14 days
  Triglyceride was analysed with Randox kit and measured in mg/dL on the 14th day
Change from Baseline Triglyceride on the 28th day | 28 days
  Triglyceride was analysed with Randox kit and measured in mg/dL on the 28th day
Change from Baseline High Density Lipoprotein Cholesterol on the 14th day | 14 days
  High Density Lipoprotein Cholesterol was analysed with Randox kit and measured in mg/dL on the 14th day
Change from Baseline High Density Lipoprotein Cholesterol on the 28th day | 28 days
  High Density Lipoprotein Cholesterol was analysed with Randox kit and measured in mg/dL on the 28th day
Change from Baseline Low Density Lipoprotein Cholesterol on the 14th day | 14 days
  Low Density Lipoprotein Cholesterol was analysed with Randox kit and measured in mg/dL on the 14th day
Change from Baseline Low Density Lipoprotein Cholesterol on the 28th day | 28 days
  Low Density Lipoprotein Cholesterol was analysed with Randox kit and measured in mg/dL on the 28th day
Change form Baseline Alanine Aminotransferase on the 14th day | 14 days
  Alanine aminotransferase was analysed with Randox kit and measured in U/L on the 14th day
Change form Baseline Alanine Aminotransferase on the 28th day | 28 days
  Alanine aminotransferase was analysed with Randox kit and measured in U/L on the 28th day
Change form Baseline Aspartate Aminotransferase on the 14th day | 14 days
  Aspartate aminotransferase was analysed with Randox kit and measured in U/L on the 14th day
Change form Baseline Aspartate Aminotransferase on the 28th day | 28 days
  Aspartate aminotransferase was analysed with Randox kit and measured in U/L on the 28th day
Change form Baseline Blood Urea Nitrogen on the 14th day | 14 days
  Blood Urea Nitrogen was analysed with Randox kit and measured in mg/dL on the 14th day
Change form Baseline Blood Urea Nitrogen on the 28th day | 28 days
  Blood Urea Nitrogen was analysed with Randox kit and measured in mg/dL on the 28th day
Change form Baseline Serum Creatinine on the 14th day | 14 days
  Serum Creatinine was analysed with Randox kit and measured in mg/dL on the 14th day
Change form Baseline Serum Creatinine on the 28th day | 28 days
  Serum Creatinine was analysed with Randox kit and measured in mg/dL on the 28th day
Change form Baseline Albumin on the 14th day | 14 days
  Albumin was analysed with Randox kit and measured in g/dL on the 14th day
Change form Baseline Albumin on the 28th day | 28 days
  Albumin was analysed with Randox kit and measured in g/dL on the 28th day
Change form Baseline Hematocrit on the 14th day | 14 days
  Hematocrit was analysed in the laboratory and measured in % on the 14th day
Change form Baseline Hematocrit on the 28th day | 28 days
  Hematocrit was analysed in the laboratory and measured in % on the 28th day
Change form Baseline Hemoglobin on the 14th day | 14 days
  Hemoglobin was analysed in the laboratory and measured in g/dL on the 14th day
Change form Baseline Hemoglobin on the 28th day | 28 days
  Hemoglobin was analysed in the laboratory and measured in g/dL on the 28th day
Change form Baseline White Blood Cell count on the 14th day | 14 days
  White Blood Cell counts was analysed in the laboratory and measured in 10*3/ µL on the 14th day
Change form Baseline White Blood Cell count on the 28th day | 28 days
  White Blood Cell counts was analysed in the laboratory and measured in 10*3/ µL on the 28th day
Change form Baseline Total Protein on the 14th day | 14 days
  Total Protein was analysed in the laboratory and measured in g/dL on the 14th day
Change form Baseline Total Protein on the 28th day | 28 days
  Total Protein was analysed in the laboratory and measured in g/dL on the 28th day
Change form Baseline Pulse on the 14th day | 14 days
  Pulse was measured with the BP monitor in /min on the 14th day
Change form Baseline Pulse on the 28th day | 28 days
  Pulse was measured with the BP monitor in /min on the 28th day

SECONDARY OUTCOMES:
Change from Baseline Body Mass Index on the 14th day | 14 day
  Body mass index measure in kg/sq m was calculated from a measure of weight in kg and height in meters on the 14 day
Change from Baseline Body Mass Index on the 28th day | 28 day
  Body mass index measure in kg/sq m was calculated from a measure of weight in kg and height in meters on the 14 day

CONTACTS AND LOCATIONS:
Overall Officials: Segun J Showande, Ph.D, Principal Investigator — University of Ibadan
Locations (1):
- Department of Clinical Pharmacy Laboratory, University of Ibadan, Ibadan, Oyo State, Nigeria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pattanittum P, Ngamjarus C, Buttramee F, Somboonporn C. Roselle for hypertension in adults. Cochrane Database Syst Rev. 2021 Nov 27;11(11):CD007894. doi: 10.1002/14651858.CD007894.pub3. PMID 34837382